CLINICAL TRIAL: NCT03676205
Title: Randomized Clinical Trial About the Therapeutic Use of Platelet-Rich Plasma (PRP) for the Treatment of Acute Muscular Injuries in Football Players.
Brief Title: Platelet-Rich Plasma in Acute Muscle Injuries
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Principal Investigator, Javier González Iglesias, Medical Doctor (orthopedic surgeon), University of the Basque Country (UPV/EHU)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRP-MUSCULO-2014-2019
Record Dates: First submitted 2018-09-13; First posted 2018-09-18 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Muscle Injury
Keywords: Platelet-Rich Plasma; hamstrings; cuadriceps; football players
MeSH Terms: interventions — Traumeel S

STUDY DESIGN:
Intervention Model Description: Two homogeneus groups with 1:1 possibilities to receive PRP or a homeopathic product.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient doesn't know the treatment. The person who analyze the data (outcomes assessor) doesn't know the treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet-Rich Plasma (Experimental): 24-72 hours after having a muscular lesion, the doctor injects an intramuscular ecoguided infiltration of 6-7 ml of PRP .
  After 4-5 days from the injury the patient starts physiotherapy adapted by stages, according to the muscular group affected.
  After 7 days from the first infiltration, the patient will recived the second infiltration of 6-7 ml of PRP.
  Interventions: Biological: PRP
- Traumel ® (Other): 24-72 hours after having a muscular lesion, the doctor injects an intramuscular ecoguided infiltration of 4 ml of a homeopathic product (Traumeel ®) After 4-5 days from the date of injury, the patient starts physiotherapy adapted by stages, according to the muscular group affected.
  After 7 days from the first infiltration, the patient will receive the second infiltration of 4 ml of a homeopathic product.
  Interventions: Other: Traumeel

INTERVENTIONS:
Biological: PRP — Platelet-Rich Plasma
  Arms: Platelet-Rich Plasma
Other: Traumeel — Homeophatic Treatment
  Arms: Traumel ®

SUMMARY:
OBJECTIVE: To evaluate the effect of Platelet Rich Plasma (PRP) injection in muscle injuries. The investigators check football players in the acute phase of hamstrings or quadriceps injuries.

Efficacy and safety are evaluated. There are two intramuscular infiltration of PRP (Ortho pras ® system) or a homeopathic product (Traumeel ®) in each of the football players. The number of days between the date of injury and the return to play, the pain, the recurrence and the adverse reactions are registered.

DETAILED DESCRIPTION:
STUDY DESIGN: Randomized Clinical Trial.

METHODS:

41 football players are included in the study. It is used randomly PRP injection or a homeopathic product in muscle injuries (hamstring), in the early stage (first 48-72 hours).

One week later, the investigators do a second infiltration with the same product, always ultrasound guided. 3-4 weeks after the injury, different variables are evaluated: the injurie with ultrasounds , self-perception test, muscle strength, flexibility, jump and run. It is compared the elapsed time in days in each of the groups: RETURN TO PLAY.

Furthermore, the PAIN, RECURRENCE RATE and ADVERSE REACTIONS are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old.
* Acute muscular Injury Type 3a-3b (Múnich classification) in hamstring muscles
* Informed consent signed

Exclusion Criteria:

* Hamstring injury (last 6 months).
* Previous infiltration in hamstring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2020-01-08 (Actual)

PRIMARY OUTCOMES:
Return to play (recovery period) | average of 3-6 weeks. Until play again a football match (training or competition)
  Days elapsed since muscular injury apperars until the return to play
Pain intensity | 3 months since the injury
  Pain after the muscle injury, and after the injections, with:
  -Funtional outcomes: pain (0 no pain; 10 unbearable pain) at rest, walking and going up and down the stairs.
  The Brief Pain Inventory - Short Form. Pain intensity (0, no pain - 10 unbearable) and interferences with the daily activities (0, does not interfere; 10, completely interferes).

SECONDARY OUTCOMES:
Incidence of Recurrences | Less than 6 months since the first injury
  Recurrence: other injury in the same muscle group during the 6 months after the first injury Complication: other injurie or disease in other location of the body (no in the same muscular group).
Number of adverse effects | Through study completion, an average of 1 year
  Any reaction with the product injected

CONTACTS AND LOCATIONS:
Overall Officials: Javier Gonzalez Iglesias, Dr, Principal Investigator — Basque Health System - Osakidetza
Locations (1):
- Javier Gonzalez Iglesias, Bilbao, Bizkaia, Spain

REFERENCES:
- [Result] Gonzalez-Iglesias J. [Therapeutic potential of platelet rich plasma. Reflections on its research and development]. Rev Esp Cir Ortop Traumatol. 2013 Jul-Aug;57(4):237-9. doi: 10.1016/j.recot.2013.04.001. Epub 2013 May 28. No abstract available. Spanish. PMID 23885648